CLINICAL TRIAL: NCT02464059
Title: Cathelicidin and Vitamin D: Impact on Populations At-Risk and With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-2200
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Cathelicidin; Vitamin D
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): Oral supplementation with 50,000 IU vitamin D3 weekly for eight weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Oral supplementation with 50,000 IU vitamin D3 weekly for eight weeks in individuals with reduced vitamin D levels.
  Other Names: cholecalciferol

SUMMARY:
This proposal will evaluate a potential mechanism of increased risk of lung function impairment, cathelicidin levels, as well as determine if vitamin D replacement can alter this pathway. This study will improve the understanding of factors which can lead to chronic lung disease. If effective, this application would also provide the justification to study vitamin D as a therapy to improve lung health.

DETAILED DESCRIPTION:
Understanding mechanisms leading to decrements in lung function, the physiologic hallmark of obstructive lung diseases including chronic obstructive pulmonary disease (COPD), are necessary to inform interventions to improve lung health. The antimicrobial peptide cathelicidin, and its primary regulator vitamin D, has been implicated in development and progression of chronic lung disease. In this study, the investigators will evaluate the effect of oral vitamin D supplementation on lung cathelicidin levels in humans. Cathelicidin has bactericidal and inflammatory activities in the lung and is regulated by vitamin D levels. The investigators hypothesize that oral vitamin D supplementation will raise cathelicidin levels in the pulmonary compartment, thereby restoring lung cathelicidin deficiency. To test this hypothesis, the investigators will recruit from two ongoing cohort studies: 1) At Johns Hopkins, the Subpopulations and Intermediate Outcome Measures in COPD Study study and 2)at University of North Carolina at Chapel Hill pulmonary and general medicine clinic. The investigators will measure blood and lung lavage cathelicidin levels in 40 vitamin D insufficient individuals (20 from each cohort) before and after eight weeks of oral vitamin D supplementation to determine the effect of vitamin D supplementation on cathelicidin levels.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65 who are current or former smokers
* Serum calcium<10.5mg/dL
* 25-Hydroxy Vitamin D (OHD)<20 ng/mL
* Creatinine Clearance ≥60 mL/min as estimated by the Cockcroft-Gault equation
* Women of reproductive potential with negative serum or urine pregnancy test and subjects must refrain from participating in a conception process and subject/partner must use at least 2 reliable forms of contraceptives for the duration of the study
* For participants with COPD, Forced Expiratory Volume in 1 second (FEV1) greater than 50% predicted.
* For smokers, current cigarette use (defined as regularly smoking 5 cigarettes per day)

Exclusion Criteria:

* Current use of vitamin D supplements
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations
* Pregnancy or currently breast-feeding
* History of nephrolithiasis
* HIV positive serostatus
* Continuous oxygen use >2 liters/min via nasal cannula
* Any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Drummond, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Johns Hopkins Clinical Research Unit, Baltimore, Maryland
  - Meadowmont Pulmonary Research Clinic, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 11/10/2015-11/15/2018
Period: Overall Study
Arm/Group | Vitamin D3
Started | 23
Completed | 17
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D3
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lung Cathelicidin Level at 8 Weeks
Description: Change from baseline to 8 weeks in bronchoscopic lavage lung cathelicidin levels after vitamin D supplementation (comparison between pre- and post-supplementation cathelicidin levels using paired t-tests for repeated measures)
Time Frame: Baseline and 8 weeks
Population: Analysis population represents N=17 participants who completed all study procedures
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Vitamin D3
Number analyzed (Participants) | 17
pg/mL | -65.5 [-172.4 to 41.3]
Statistical Analysis 1: Comparison: Vitamin D3; Test type: Superiority; p = 0.21, t-test, 2 sided — P-value is not adjusted for multiple comparisons. A priori threshold for significance is p<0.05; Mean Difference (Final Values) = -65.5, 95% CI 2-sided [-172.4 to 41.3], Standard Deviation 207.8

2. Secondary Outcome: Change From Baseline in Blood Cathelicidin at 8 Weeks
Description: Change from baseline to 8 weeks in blood cathelicidin levels after vitamin D supplementation (comparison between pre- and post-supplementation cathelicidin levels using paired t-tests for repeated measures)
Time Frame: Baseline and 8 weeks
Population: Analysis population represents N=17 participants who completed all study procedures
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D3
Number analyzed (Participants) | 17
ng/ml | -0.55 (12.6)
Statistical Analysis 1: Comparison: Vitamin D3; Test type: Superiority; p = 0.86, t-test, 2 sided — P-value is not adjusted for multiple comparisons. A priori threshold for significance is p<0.05; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-7.02 to 5.91], Standard Deviation 12.6

3. Secondary Outcome: Change From Baseline in Blood Vitamin D Binding Protein at 8 Weeks
Description: Change from baseline to 8 weeks in blood vitamin D binding protein after vitamin D supplementation (comparison between pre- and post-supplementation cathelicidin levels using paired t-tests for repeated measures)
Time Frame: Baseline and 8 weeks
Population: The outcome measure of Vitamin D Binding Protein was not collected nor assessed on any study participants. This was due to technical limitations related to the assay.
Arm/Group | Vitamin D3
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of informed consent until final bronchoscopy procedure, an approximate total of 8 weeks.
Arm/Group | Vitamin D3
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 (N=23)
Death after house fire (General disorders) | 1 (1) — Participant was involved in house fire while on study.

LIMITATIONS AND CAVEATS:
Study enrollment did not achieve targeted sample size enrollment during the time frame of the funding award.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT02464059/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT02464059/SAP_001.pdf